CLINICAL TRIAL: NCT06912490
Title: Proteomic Analysis of Amniotic Fluid to Predict Postnatal Renal Function in Fetuses With Renal and Urinary Tract Malformations
Acronym: PAPER FACE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/24/0291; ID-RCB : 2024-A01612-45 (Other: ANSM)
Record Dates: First submitted 2025-03-21; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Kidney Diseases
Keywords: Antenatal; fetal bilateral nephropathies; renal function; prognosis; proteomic analysis; renal ultrasound
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Proteomic-Based Prediction of Postnatal Kidney Function in Fetuses with Bilateral CAKUT (Experimental)
  Interventions: Other: Amniotic Fluid Proteomic Analysis Using Capillary Electrophoresis-Mass Spectrometry (CE-MS)

INTERVENTIONS:
Other: Amniotic Fluid Proteomic Analysis Using Capillary Electrophoresis-Mass Spectrometry (CE-MS) — This intervention consists of analyzing the amniotic fluid proteome using capillary electrophoresis coupled with mass spectrometry (CE-MS). The goal is to evaluate a predefined 98-peptide signature that predicts postnatal kidney function in fetuses with bilateral congenital anomalies of the kidney and urinary tract. Unlike standard prenatal assessments based on ultrasound and fetal biochemistry, this method provides a molecular-based prognostic tool to improve decision-making regarding pregnancy management and neonatal care

SUMMARY:
The aim of this project is to validate a previously established amniotic fluid 98 peptide signature predictive of post-natal outcome in fetuses with congenital anomalies of the kidney and the urinary tract (CAKUT) in a "real" clinical context. It includes the feasibility of collecting, transporting and analyzing the amniotic fluid peptidome from clinical centers all over France and of providing the result in a clinically accepted time-frame. Therefore, this multicenter study will not only allow to determine the added value of such new prenatal test but also to ensure the feasibility of its introduction in the management of CAKUT pregnancies.

DETAILED DESCRIPTION:
CAKUT represent 20-30% of all inborn malformations. Whereas prognosis is generally favorable in unilateral disease, bilateral CAKUT are the predominant causes of chronic kidney disease (CKD) in childhood and account for ~50% of pediatric and young adult end stage renal disease (ESRD) cases. Current ultrasound- or amniotic fluid biochemistry-based prenatal clinical advice to parents expecting a child with bilateral CAKUT is far from accurate. This prognostic uncertainty of disease progression has particularly serious implications for parents confronted with the decision of continuation or elective termination of pregnancy. Such uncertainty has led to documented situations where half of the cases of severe bilateral CAKUT for whom termination of pregnancy was considered but not performed had normal postnatal renal function. In the case parents decide to continue the pregnancy, knowledge of the precise outcome would allow anticipating dialysis, transplantation or palliative care. 98 peptide signature have been identified in amniotic liquid that predicted with high sensitivity and specificity postnatal kidney function in fetuses with CAKUT (Klein, Buffin-Meyer et al., Kidney Int 2021).

The aim of the current project is to validate this signature in an independent multicenter French study and determine added value and feasibility of its introduction in the routine management of CAKUT pregnancies.

After the discovery of a CAKUT pregnancy in an associated French center and approval and informed consent of the parents, part of the amniotic fluid (~ 1 mL) that is routinely collected for chromosomal anomalies is transferred to the research laboratory Inserm U1297 in Toulouse. The peptide content of the amniotic fluid is analyzed allowing the evaluation of the abundance of the 98 peptides of the signature. It will result in a risk score for developing severe kidney failure before the age of 2 years, postnatally. This score will be communicated by the clinicians from Toulouse responsible for the project to the clinicians of the center requesting the analysis.

ELIGIBILITY:
Inclusion Criteria:

* All fetuses with bilateral renal development anomalies with structural changes in the parenchyma, with or without associated urinary tract anomalies;
* Signed informed consent of the mother
* Non-opposition of the father.

Exclusion Criteria:

* Unilateral abnormality of renal development
* Any pregnancy for which amniocentesis may represent a risk for the fetus or the mother
* Twin pregnancies
* Pregnant woman protected by law (guardianship, curatorship)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2029-12-20 (Estimated); Study Completion 2029-12-20 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the test in the evaluation of renal survival (need for dialysis) and patient survival at 2 years of life. | 2 years of age
  Renal survival is defined as the absence of end-stage renal disease (ESRD) requiring dialysis by 2 years of age. Patient survival is defined as the child being alive at 2 years. Renal function is assessed through clinical follow-up, including serum creatinine measurements and estimated glomerular filtration rate (eGFR) using the Schwartz formula. Dialysis initiation is determined based on standard clinical criteria for ESRD. Survival status is confirmed through medical records and follow-up visits. This outcome aims to validate the predictive value of the 98-peptide amniotic fluid signature for postnatal kidney function in CAKUT fetuses.

SECONDARY OUTCOMES:
Sensitivity and specificity of the test in the evaluation of postnatal renal function estimated by the Schwartz formula and his serum creatinine | At months 1, 6, 12, and 24 postnatally
  Schwartz formula which is based on the patient's height (T, in cm) and his serum creatinine (Creat, in µmol/L) (T*36.5/Creat)
Severity score result rendering time | up to 2 weeks after sample collection
  measure of the delay to give the result to the investigator site

CONTACTS AND LOCATIONS:
Locations (1):
- Children Hospital, Toulouse, France